CLINICAL TRIAL: NCT07307222
Title: Effect of Transcutaneous Tibial Nerve Stimulation on Primary Dysmenorrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Atef Mahmoud Sonbol, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005880
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard physical therapy program (Active Comparator): It will include 18 females with primary dysmenorrhea who will receive standard physical therapy program for 3 months. Hot pack or heating pad will be applied to the lower abdomen or lower back area for 15-20 minutes per session, with 3 sessions per week over a period of 12 weeks. Six stretching exercises will be applied.The females will be instructed to perform the exercise 3 days/week.
  Interventions: Other: Standard physical therapy program
- Standard physical therapy program + Transcutaneous Tibial Nerve Stimulation (TTNS) (Experimental): It will include 18 females with primary dysmenorrhea who will receive TTNS 30 minutes once a week for 12 weeks, in addition to the same physical therapy program.
  Interventions: Other: Standard physical therapy program; Other: Transcutaneous Tibial Nerve Stimulation (TTNS)

INTERVENTIONS:
Other: Standard physical therapy program — The standard physical therapy program will include the application of a hot pack or heating pad to the lower abdomen or lower back for 15-20 minutes per session, three times per week for a duration of 12 weeks. The temperature of the hot pack will be maintained between 40°C and 45°C (104°F-113°F). In addition, participants will perform six stretching exercises for 30-45 minutes per session, also three times per week for 12 weeks.
Other: Transcutaneous Tibial Nerve Stimulation (TTNS) — The TTNS intervention will be applied once a week for 30-minute sessions over 12 weeks. The EV-906 electrostimulation device will be used for the treatment. A symmetrical biphasic current will be applied in continuous mode at 20 Hz and 200 μs. The patient will be in a supine position with knees flexed and abducted at a 90-degree angle. Stimulation will be applied to both legs using two adhesive electrodes placed cranially to the internal malleolus of each leg, with additional electrodes placed at the ipsilateral calcaneus. The stimulation intensity will be regulated between 1 and 30 mA.
  Arms: Standard physical therapy program + Transcutaneous Tibial Nerve Stimulation (TTNS)

SUMMARY:
This study will be conducted to evaluate the effect of Transcutaneous Tibial Nerve Stimulation (TTNS) on primary dysmenorrhea.

DETAILED DESCRIPTION:
Primary dysmenorrhea is a common, disregarded, underdiagnosed, and inadequately treated complaint of both young and adult females. It negatively impacts the quality of life of young females, forming the main reason behind their absenteeism from school or work, and causing limitation of daily activities and psychological stress.

The Transcutaneous Tibial Nerve Stimulation (TTNS) is a rather new method acclaimed to be viable for chronic pelvic pain management. As it uses surface electrodes, it can be self-administrated by patients. Research is lacking regarding the effect of TTNS on primary dysmenorrhea. Thus, this study will be designed to examine the effect of TTNS on menstrual pain and distress as well as quality of life in females with primary dysmenorrhea. Study results will have valuable benefits in the physical therapy field, scientific research and medical and health organizations.

ELIGIBILITY:
Inclusion Criteria:

* Females with a regular menstrual cycle, experiencing primary dysmenorrhea, confirmed by history and clinical diagnosis.
* Females aged between 18 and 35 years.
* Their BMI ranging from 20 to 29.9 kg/m².

Exclusion Criteria:

* Females engaging in regular physical exercises prior to the study course.
* A history of abdominal or pelvic surgery.
* Pelvic pathologies or diseases (e.g., polycystic ovary syndrome, endometriosis, adenomyomas, or uterine fibroids).
* Malignant or benign neoplasms in the uterus.
* Chronic diseases, including diabetes and/or rheumatoid arthritis.
* Presence of metal implants or pacemakers.
* Any contraindications to the use of electrical stimulation (e.g., open wounds, some skin conditions…. etc.).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-21 (Estimated); Primary Completion 2026-03-21 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Menstrual pain intensity | 3 months
  Using the Visual Analog Scale (VAS), each female will be asked to rate her menstrual pain intensity by placing a mark along the line that corresponds to their perceived pain level now. The distance from the "no pain" end to the female's mark will be then measured in centimeters to quantify the pain intensity. A higher value indicates greater pain intensity.
Assessment of Menstrual Distress | 3 months
  Using the Menstrual Distress Questionnaire (MEDI-Q), each participant will report physical, emotional, and social symptoms experienced during menstruation over the past 12 months and rate their impact on daily functioning and quality of life. The questionnaire uses a Likert scale to evaluate symptoms from the most recent cycle, and a total score is obtained by summing responses. Higher scores indicate greater menstrual distress and more substantial psychological and physical effects.
Assessment of Menstrual symptoms | 3 months
  Using the WaLIDD score, each female will be asked to answer questions by putting a score regarding five key factors related to primary dysmenorrhea: Working ability, Location of pain, Intensity of pain, Days of pain, and the presence of Dysmenorrhea. Each factor is scored based on the female's experience during their menstrual cycle. The scores from all factors are combined to produce a total score, with a higher score indicating greater severity and impact of dysmenorrhea.

SECONDARY OUTCOMES:
Assessment of Quality of Life | 3 months
  The World Health Organization Quality of Life (WHOQOL-26) questionnaire will be used to assess each participant's perceived quality of life, health, and daily functioning. Participants answer all items and are advised to select the response that feels most appropriate, often their first instinct. Scores for the four domains-physical, psychological, social, and environmental-are averaged to produce an overall score. Higher scores indicate better quality of life, while lower scores reflect greater impairment. This tool helps evaluate how conditions such as dysmenorrhea affect overall well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Afaf Mohamed Botla, PhD, Study Chair — Assistant Professor, Cairo University; Hossam Eldeen Hussein Kamel, PhD, Study Director — Professor, Al-Azhar university; Mahitab Mohamed Yosri Ibrahim, PhD, Study Director — Lecturer, Cairo university
Locations (1):
- Damas Central Hospital, Al Mansurah, Egypt